CLINICAL TRIAL: NCT05368285
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Dose-finding Study to Assess the Efficacy and Safety of CDX-0159 in Patients With Chronic Spontaneous Urticaria
Brief Title: A Phase 2 Study of CDX-0159 in Patients With Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-06; 2021-006413-11 (EudraCT Number)
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CDX-0159; barzolvolimab
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- barzolvolimab 75 mg then 150 mg (Experimental): barzolvolimab 75 mg injection subcutaneous every 4 weeks for 16 weeks and then 150 mg injection subcutaneous every 4 weeks for 36 weeks
  Interventions: Biological: barzolvolimab
- barzolvolimab 75 mg then 300 mg (Experimental): barzolvolimab 75 mg injection subcutaneous every 4 weeks for 16 weeks and then 300 mg injection subcutaneous every 8 weeks for 36 weeks
  Interventions: Biological: barzolvolimab
- barzolvolimab 150 mg (Experimental): barzolvolimab 150 mg injection subcutaneous every 4 weeks for 52 weeks
  Interventions: Biological: barzolvolimab
- barzolvolimab 300 mg (Experimental): barzolvolimab 300 mg injection subcutaneous every 8 weeks for 52 weeks
  Interventions: Biological: barzolvolimab
- Placebo then barzolvolimab 150 mg (Experimental): Placebo injection subcutaneous every 4 weeks for 16 weeks and then barzolvolimab 150 mg injection subcutaneous every 4 weeks for 36 weeks
  Interventions: Biological: barzolvolimab; Drug: Matching Placebo
- Placebo then barzolvolimab 300 mg (Experimental): Placebo injection subcutaneous every 4 weeks for 16 weeks and then barzolvolimab 300 mg injection subcutaneous every 8 weeks for 36 weeks
  Interventions: Biological: barzolvolimab; Drug: Matching Placebo

INTERVENTIONS:
Biological: barzolvolimab — Subcutaneous Administration
  Other Names: CDX-0159
Drug: Matching Placebo — Subcutaneous Administration
  Arms: Placebo then barzolvolimab 150 mg; Placebo then barzolvolimab 300 mg

SUMMARY:
The purpose of this study is to assess the clinical effect, the pharmacodynamics, the safety, and the pharmacokinetics of barzolvolimab (CDX-0159) in patients with Chronic Spontaneous Urticaria

DETAILED DESCRIPTION:
The purpose of this study is to assess the clinical effect, the pharmacodynamics, the safety, and the pharmacokinetics of barzolvolimab in patients with Chronic Spontaneous Urticaria.

There is a screening period of up to 4 weeks, followed by a 16-week placebo-controlled treatment period (Placebo-Controlled Treatment Phase) where patients will receive either barzolvolimab at a dose level of 75mg, 150mg, or 300mg, or placebo, and then a 36-week treatment period where all patients will receive barzolvolimab. Patients who receive barzolvolimab 75mg or placebo in the placebo-controlled treatment phase will be re-randomized to receive either barzolvolimab 150mg or 300mg in the active treatment phase.

ELIGIBILITY:
Key inclusion criteria:

1. Males and females, >/= 18 years of age.
2. Diagnosis of chronic spontaneous urticaria (CSU) >/= 6 months.
3. Diagnosis of CSU despite the use of a stable regimen of second generation non-sedating H1-antihistamine as defined by:

   1. The presence of hives for >/= 6 weeks at any time prior to Visit 1 despite the use of H1-antihistamines.
   2. Must be on a stable regimen of second generation non-sedating H1-antihistamine for >/= 4 weeks prior to study treatment.
   3. UAS7 of >/= 16 and ISS7 of >/= 8 during the 7 days prior to treatment.
4. Normal blood counts and liver function tests
5. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days after treatment.
6. Willing and able to complete a daily symptom electronic diary and comply with study visits.

Key exclusion criteria:

1. Women who are pregnant or nursing.
2. Clearly defined cause for chronic urticaria.
3. Active, pruritic skin condition in addition to CSU.
4. Medical condition that would cause additional risk or interfere with study procedures.
5. Known active HIV, hepatitis B or hepatitis C infection.
6. Vaccination of a live vaccine within 2 months prior to study treatment (subjects must agree to avoid vaccination during the study). Inactivated vaccines are allowed such as seasonal influenza injection or COVID-19 vaccine.
7. History of anaphylaxis
8. Prior treatment with barzolvolimab

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to Week 12 of UAS7 (Urticaria Activity Score) | From baseline to Day 85 (Week 12)
  Evaluate efficacy of barzolvolimab on urticaria activity as measured by urticaria activity score (UAS). UAS7 is the sum of the itch severity score measured over 7 days (ISS7) and the hives severity score measured over 7 days (HSS7). The possible range of UAS7 is 0 - 42.
  Itch severity score (ISS) is on a scale of 0 - 3.
  0 = None
  1. = mild (present, but not annoying or troublesome)
  2. = moderate (troublesome, but does not interfere with normal daily activity or sleep)
  3. = intense (severe itch, which is sufficiently troublesome to interfere with normal daily activity or sleep)
  Hives severity score (HSS) is on a scale of 0 - 3.
  0 = None
  1. = less than 20 hives
  2. = between 20 and 50 hives
  3. = greater than 50 hives

SECONDARY OUTCOMES:
Mean change from baseline to Week 12 of ISS7 (Itch Severity Score) | From baseline to Day 85 (Week 12)
  ISS7 is derived by adding up the daily scores over 7 days. The possible range of the weekly score is 0 -21.
Mean change from baseline to Week 12 of HSS7 (Hives Severity Score) | From baseline to Day 85 (Week 12)
  HSS7 is derived by adding up the daily scores over 7 days. The possible range of the weekly score is 0 -21.
Mean change from baseline to Week 12 of AAS7 (Angioedema Activity Score) | From baseline to Day 85 (Week 12)
  AAS captures the presences of swelling over the last 24 hours and rates the severity with 5 questions. The possible range of the weekly score is 0 - 105.

CONTACTS AND LOCATIONS:
Locations (56):
- United States (13):
  - Clinical Research Center of Alabama dba Allervie Clinical Research, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - Little Rock Allergy & Asthma CRC, Little Rock, Arkansas
  - Kern Research, Inc, Bakersfield, California
  - Allergy & Asthma Consultants, Redwood City, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Treasure Valley Medical Research, Boise, Idaho
  - Allergy & Asthma Specialists, PSC, Owensboro, Kentucky
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Chesapeake Clinical Research, White Marsh, Maryland
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center/Subspeciality-Allergy and Immunology, The Bronx, New York
- Bulgaria (5):
  - "Diagnostic Consultative Center Pulmed" EOOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv
  - Outpatient clinic for individual practice for specialized outpatient medical care in allergology-Doctor Thalat Sally Cholak EOOD, Razgrad
  - Medical Center Iskar EOOD Office of Clinical Allergology, Sofia
  - Medical Center "SYNEXUS SOFIA", EOOD, Sofia
- Vahlberg & Pild Clinic, Tallinn, Estonia
- Georgia (3):
  - Healthy Future, Tbilisi
  - Center of Allergy and Immunology, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (10):
  - LMU Klinikum - Klinik und Poliklinik für Dermatologie und Allergologie DASZ-Dermato-Allergologisches Studien Zentrum, München, Bavaria
  - Universitaetsklinikum Giessen u. Marburg GmbH, Marburg, Hesse
  - Hannover Medical University, Hanover, Lower Saxony
  - Klinikum Oldenburg gGmbH - Klinik f. Dermatologie u. Allergologie, Oldenburg, Lower Saxony
  - Universitätsklinikum Düsseldorf - Dermatologie, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Münster Klinik u. Poliklinik f. Dermatologie, Münster, North Rhine-Westphalia
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein - Zentrum für entzündliche Hauterkrankunge, Kiel, Schleswig-Holstein
  - Charite - Institute of Allergology IFA Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Heidelberg - Dermatologie, Heidelberg
- Hungary (4):
  - Semmelweis Egyetem, ÁOK, Bőr-, Nemikórtani és Bőronkológiai Klinika, Budapest
  - Debreceni Egyetem, ÁOK és KK, Bőrgyógyászati Tanszék és Bőrgyógyászati Klinika, Debrecen
  - Allergo-Derm Bakos Kft. Bőrgyógyászati Magánrendelő, Szolnok
  - Óbudai Egészségügyi Centrum Kft., Zalaegerszeg
- Poland (8):
  - Centrum Medyczne Plejady, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 w Lodzi, Lodz
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Prof. Doroty Krasowskie, Lublin
  - Uniwersytecki Szpital Kliniczny w Opolu, Pododdział Chorób Wewnętrznych i Alergologii, Opole
  - Medicome Sp. z o.o., Oświęcim
  - Medicover Integrated Clinical Services Sp. Z.o.o., Torun
  - Klinika Ambroziak sp. z o.o., Warsaw
- South Africa (8):
  - Iatros International, Bloemfontein, Free State
  - WorthWhile Clinical Trials, Benoni, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Ubuntu Clinical Research, Lenasia, Gauteng
  - FCRN Clinical Trial Centre Vaal Triangle, Vereeniging, Gauteng
  - Synapta Clinical Research, Durban, KwaZulu-Natal
  - Dr Pj Sebastian, Durban, KwaZulu-Natal
  - The University of Cape Town - Lung Institute, Cape Town
- Spain (4):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Bellvitge, Barcelona
  - Universidad de Navarra, Madrid